CLINICAL TRIAL: NCT06574828
Title: A Randomized, Double-Blind, Placebo- and Positive-Controlled (Moxifloxacin), Parallel Study With a Nested Crossover to Assess the Effect of Multiple Oral Therapeutic and Supratherapeutic Doses of BIIB091 on Cardiac Repolarization in Healthy Participants
Brief Title: A Study to Find Out How Multiple Doses of BIIB091 Affect the Electrical Activity of the Heart in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 257HV109
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — BIIB091; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BIIB091, BIIB091-matched placebo, Moxifloxacin-matched placebo (Experimental): Participants will receive BIIB091, BIIB091-matched placebo, and moxifloxacin-matched placebo orally during the inpatient period (Days -1 to 13).
  Interventions: Drug: BIIB091; Drug: BIIB091-matched Placebo; Drug: Moxifloxacin-matched Placebo
- Moxifloxacin, Moxifloxacin-matched placebo, BIIB091-matched placebo (Active Comparator): Participants will receive moxifloxacin, moxifloxacin-matched placebo, and BIIB091-matched placebo orally during the inpatient period (Days -1 to 13).
  Interventions: Drug: Moxifloxacin; Drug: BIIB091-matched Placebo; Drug: Moxifloxacin-matched Placebo

INTERVENTIONS:
Drug: BIIB091 — Administered as specified in the treatment arm.
  Arms: BIIB091, BIIB091-matched placebo, Moxifloxacin-matched placebo
Drug: Moxifloxacin — Administered as specified in the treatment arm.
  Arms: Moxifloxacin, Moxifloxacin-matched placebo, BIIB091-matched placebo
Drug: BIIB091-matched Placebo — Administered as specified in the treatment arm.
Drug: Moxifloxacin-matched Placebo — Administered as specified in the treatment arm.

SUMMARY:
In this study, researchers will learn how the heart reacts to multiple doses of BIIB091 in healthy participants. In previous studies looking at BIIB091, researchers have found that a certain range of doses can cause changes in the electrical activity of the heart. In this study, researchers want to learn more about that activity after participants take BIIB091 at lower and higher doses for 5 days. The main objective of this study is to learn how the heart's electrical activity changes after taking BIIB091. To measure this, researchers will look at something called the QT interval corrected for heartbeat, also known as "QTc". This represents the time it takes for the heart to contract and relax. A QT interval that is too long means that the heart's electrical system is taking longer than normal to recharge between heartbeats. This could increase the risk of abnormal heartbeats that may lead to sudden death.

The main questions researchers want to answer are:

• What is the change in the participants' QTc after taking BIIB091?

Researchers will also learn more about:

* Any changes in other measures of the heart's electrical activity
* How the body processes BIIB091, as well as something called "M23", which is made in the body when BIIB091 is broken down
* Any medical problems the participants have during the study
* Any changes in the participants' overall health during the study

This study will be done as follows:

* Participants will be screened to check if they can join the study. The screening period will be up to 29 days, after which participants will check into their study research center.
* Participants will be randomly assigned to be in 1 of 2 groups:

  * Group 1: Participants will take a low dose of BIIB091 for 5 days followed by a high dose of BIIB091 for 5 days.
  * Group 2: Participants will take a single dose of moxifloxacin. Moxifloxacin is an antibiotic used to treat bacterial infections. Researchers are using it in this study to compare to BIIB091, because it is known to cause abnormal changes to the heart's electrical activity.
  * Participants in both Group 1 and Group 2 will also take a placebo while at the study research center. A placebo looks like the study drug or moxifloxacin, but does not have any real medicine in it.
* Participants will remain at their study research center for 15 days. Afterwards, there will be a follow-up visit 11 to 14 days after each participant's last dose. Each participant will be in the study for up to 57 days.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the effect of BIIB091 and its metabolite M23 following multiple therapeutic and supratherapeutic doses of BIIB091 on QTc intervals in healthy participants. The secondary objectives of this study are: to evaluate the effect of BIIB091 and its metabolite M23 following multiple therapeutic and supratherapeutic doses of BIIB091 on other electrocardiogram (ECG) parameters (heart rate [HR], pulse rate [PR] and QRS intervals, and ECG morphology); to demonstrate assay sensitivity of the study to detect a QTc effect using moxifloxacin as a positive control; to assess the pharmacokinetics (PK) of BIIB091 and its metabolite M23, following multiple oral dose administrations in healthy participants; to evaluate the safety and tolerability of BIIB091 in healthy participants.

ELIGIBILITY:
Key Inclusion criteria:

* Have a body mass index between 18 and 32 kilograms per meter square (kg/m^2), inclusive, and a total body weight > 50 kg, at screening and Day -2.
* Must be in good health as determined by the Investigator, based on medical history and Screening evaluations.
* Negative polymerase chain reaction (PCR) test result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at check-in (Day -2).

Key Exclusion Criteria:

* History of any clinically significant cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the Investigator.
* Clinically significant 12-lead ECG findings at screening and prior to first dose, including confirmed demonstration of QTcF > 430 milliseconds (ms), QRS > 120 ms, PR > 220 ms, or heart rate < 45 beats per minutes (bpm) based on the average of triplicate measurements, early repolarization, or any other clinically significant 12-lead ECG abnormalities as determined by the Investigator.
* History of torsades de pointes or additional risk factors for torsades de pointes.
* History of, or positive test result at Screening for, human immunodeficiency virus, hepatitis B virus, or hepatitis C virus infection.
* Use of any prescription or over-the-counter medication (including herbal supplements) that are known to prolong QT/QTc interval or induce torsades de pointes.
* Chronic, recurrent, or serious infection (e.g., pneumonia, septicemia), as determined by the Investigator, within 90 days prior to Screening or between Screening and Check-in.

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-03-22 (Actual); Study Completion 2025-03-22 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in QT Interval Corrected for Heart Rate (QTc) for BIIB091 | Baseline (Day -1) up to Day 14
Change From Baseline in QT Interval Corrected for Heart Rate (QTc) for Metabolite 23 (M23) | Baseline (Day -1) up to Day 14

SECONDARY OUTCOMES:
Change From Baseline in Heart Rate (ΔHR) for BIIB091 and M23 | Baseline (Day -1) up to Day 14
Change From Baseline in Pulse Rate Interval (ΔPR) for BIIB091 and M23 | Baseline (Day -1) up to Day 14
Change From Baseline in QRS Interval (ΔQRS) for BIIB091 and M23 | Baseline (Day -1) up to Day 14
Number of Participants With Categorical Outliers for QT Interval Corrected Formula for Heart Rate (QTcF), HR, PR, and QRS for BIIB091 and M23 | From Day -1 up to Day 14
Number of Participants With Treatment-Emergent Changes in ECG Morphology for BIIB091 and M23 | From Day -1 up to Day 14
Time to Maximum Measured Plasma Concentration (Tmax) of BIIB091 and M23 | Pre-dose and at multiple timepoints up to Day 14
Maximum Measured Plasma Concentration (Cmax) of BIIB091 and M23 | Pre-dose and at multiple timepoints up to Day 14
Area Under the Plasma Concentration Versus Time Curve to 24 Hours (AUC0-24) of BIIB091 and M23 | Pre-dose and at multiple timepoints up to Day 14
Area Under the Plasma Concentration Versus Time Curve to the Last Measurable Concentration (AUC0-t) of BIIB091 and M23 | Pre-dose and at multiple timepoints up to Day 14
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day -1 up to end of study follow-up (up to 28 days)
Number of Participants With Clinically Significant Vital Signs Abnormalities | From Day -1 up to end of study follow-up (up to 28 days)
Number of Participants With ECG Abnormalities | From Day 1 up to Day 14
Number of Participants With Clinically Significant Laboratory Assessment Abnormalities | At Days 4, 14 and follow-up (up to 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Austin Clinic PPD, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/